CLINICAL TRIAL: NCT03989843
Title: Is Cryopreserved Embryo Replacement is Associated With Higher Birthweight Compared With Fresh Embryo ? Sibling Embryo Cohort Study
Brief Title: Impact of Embryo Cryopreservation on Birth Weight
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0306
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Infertility
Keywords: ART; Birthweight; Siblings; Cryopreservation; Epigenetic; Medical assistance to procreation
MeSH Terms: conditions — Infertility; Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frozen embryo transfer: Frozen embryo transfer
- Fresh embryo transfer: Fresh embryo transfer

SUMMARY:
Birth weight (BW) is higher after frozen embryo transfer (FET) than after fresh embryo replacement. No study has compared the BW of siblings conceived using the same oocyte/embryo cohort. The aim of this study was to determine whether the freezing-thawing procedure is involved in such difference.

ELIGIBILITY:
Inclusion Criteria:

* sibling pairs where fresh embryo replacement resulting in a singleton live birth was followed by transfer of one or two frozen embryos from the same cohort that resulted in a singleton live birth, between May 2007 and June 2015.

Exclusion Criteria:

* Twin pregnancies and stillbirths were excluded. If the BW of at least one sibling was unknown, the pair was not included in the study.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: sibling pairs where fresh embryo replacement resulting in a singleton live birth was followed by transfer of one or two frozen embryos from the same cohort that resulted in a singleton live birth, between May 2007 and June 2015.
  Twin pregnancies and stillbirths were excluded. If the BW of at least one sibling was unknown, the pair was not included in the study
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2007-05-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
birthweight | 1 day
  change after FET than after fresh embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Margaux Anav, Doctor, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC